CLINICAL TRIAL: NCT07035613
Title: Investigating Chinese Herbal Medicine for Modulating Gut Microbiota in Treating Inflammatory Bowel Disease: Molecular Mechanisms and Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH113-REC2-034
Record Dates: First submitted 2025-06-08; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: IBD - Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BXD treatment (single group) (Experimental): Participants will receive BXD daily for 14 days. Plasma IgA and fecal 16S-FL sequence will be measured at baseline and after treatment.
  Interventions: Drug: BXD treatment

INTERVENTIONS:
Drug: BXD treatment — The BXD extract was obtained from Sun Ten Pharmaceutical Company and is manufactured according to the standard procedures outlined in the Taiwan Herbal Pharmacopeia IV. The extract is produced using a fixed herbal composition and ratio based on the traditional BXD formula to yield a concentrated powder. The administration of BXD in this study follows the dosage and usage guidelines specified in the Pharmacopeia.

SUMMARY:
The goal of this exploratory, single-arm intervention study is to evaluate whether Banxia Xiexin Decoction (BXD) can prevent colitis by modulating gut microbiota composition and regulating immune responses, including IgA production, in healthy adults.

The main questions it aims to answer are:

Can BXD prevent colitis by modulating gut microbiota composition? Can BXD enhance immune markers such as IgA without adverse effects?

There is no comparison group in this study.

Participants will:

Take BXD daily for 14 days. Provide stool and blood samples for microbiota analysis and immune marker testing.

Eligible participants include healthy men and women aged 20 years or older, with no major illnesses, autoimmune diseases, cancer, or recent use of antibiotics, immunosuppressants, or probiotics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged ≧20 years.
2. Participants who are able to provide signed informed consent.
3. Healthy individuals with no history of major illnesses or cancer.

Exclusion Criteria:

1. Inclusion who do not meet the inclusion criteria.
2. Individuals deemed unsuitable for participation by the investigator.
3. The individual is unable to comply with the study schedule.
4. Individuals unable to provide signed informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Changed in plasm IgA levels from baseline to Day14 measured by ELISA | From enrollment to the end for 2 time points (Day 0 and Day 14) to collect the plasma sample.
  Plasma IgA concentration will be measured at baseline (Day 0) and Day 14 using a validated ELISA method. The primary outcome will be the mean change in plasma IgA levels from baseline to Day 14.
  Time : From enrollment to Day 14

SECONDARY OUTCOMES:
Change in gut microbiota composition from baseline to Day 14 assessed by 16S rRNA full-length sequencing | Fecal samples were collected before(Day 0) and after the treatment(Day 14) period.
  Fecal samples were collected at baseline (Day 0) and on Day 14. Microbiota composition was analyzed using full-length 16S rRNA sequencing. The outcome will summarize the relative abundance of key bacteria taxa and diversity indices before and after BXD treatment.
  Time： From enrollment to Day 14.

CONTACTS AND LOCATIONS:
Locations (1):
- China medicial university hospital, Taichung, Taiwan